CLINICAL TRIAL: NCT04650087
Title: COVID-19 Post-hospital Thrombosis Prevention Trial: An Adaptive, Multicenter, Prospective, Randomized Platform Trial Evaluating the Efficacy and Safety of Antithrombotic Strategies in Patients With COVID-19 Following Hospital Discharge
Brief Title: COVID-19 Thrombosis Prevention Trials: Post-hospital Thromboprophylaxis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thomas L. Ortel (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Thomas L. Ortel, Professor, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00107078
Record Dates: First submitted 2020-11-30; First posted 2020-12-02 (Actual); Results first posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — apixaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Apixaban (Active Comparator): Drug: Apixaban 2.5 MG Participants will be given study medication at the time of discharge from the hospital. Participants will take Apixaban 2.5 MG twice a day, once in the morning and once in the evening, for 30 days. Participants will be contacted (electronic or telephone) 2 days after starting the study medication and contact will continue up to day 90 after starting study treatment. Follow up will be through electronic and/or telephone contact depending on the participant's preference, compliance, and medication adherence. Participants will be queried for any clinically relevant endpoints, especially major bleeding or a need to seek healthcare attention for any reason. Follow-up will occur from the time of discharge and through the 30 day study period, with contacts 2 days, 10 days, 20 days, and 30 days after discharge. Two additional study contacts will take place 45 days and 90 days after discharge.
  Interventions: Drug: Apixaban 2.5 MG
- Placebo (Placebo Comparator): Drug: Placebo Participants will be given study medication at the time of discharge from the hospital. Participants will take the Placebo twice a day, once in the morning and once in the evening, for 30 days. Participants will be contacted (electronic or telephone) 2 days after starting the study medication and contact will continue up to day 90 after starting study treatment. Follow up will be through electronic and/or telephone contact depending on the participant's preference, compliance, and medication adherence. Participants will be queried for any clinically relevant endpoints, especially major bleeding or a need to seek healthcare attention for any reason. Follow-up will occur from the time of discharge and through the 30 day study period, with contacts 2 days, 10 days, 20 days, and 30 days after discharge. Two additional study contacts will take place 45 days and 90 days after discharge.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apixaban 2.5 MG — Participants will take Apixaban 2.5 MG twice a day, once in the morning and once in the evening for 30 days. Participants will be contacted (electronic or telephone) 2 days after starting the study medication and will continue up to day 90 after starting study treatment. Followup will occur from the time of discharge through the 30 day study period with contacts at 2 days, 10 days, 20 days and 30 days after discharge. Two additional study contacts will take place 45 days and 90 days after discharge.
  Other Names: Eliquis
  Arms: Apixaban
Drug: Placebo — Participants will take placebo twice a day, once in the morning and once in the evening for 30 days. Participants will be contacted (electronic or telephone) 2 days after starting the study medication and will continue up to day 90 after starting study treatment. Followup will occur from the time of discharge through the 30 day study period with contacts at 2 days, 10 days, 20 days and 30 days after discharge. Two additional study contacts will take place 45 days and 90 days after discharge.
  Arms: Placebo

SUMMARY:
A multicenter, adaptive, randomized platform trial evaluating the efficacy and safety of antithrombotic strategies in patients with COVID-19 following hospital discharge

DETAILED DESCRIPTION:
This study is an adaptive, prospective, randomized platform trial designed to compare the effectiveness and safety of antithrombotic therapy with no antithrombotic therapy after hospitalization for 48 hours or longer for COVID-19. For Stage 1 of this study, participants will be randomized to either prophylactic anticoagulation or matching placebo for 30 days, and then followed for an additional 60 days after the completion of treatment (total duration of follow-up, 90 days).

The primary objective is to determine the most effective and safe antithrombotic strategy to prevent the composite outcome of symptomatic deep vein thrombosis, pulmonary embolism, other venous thromboembolism, ischemic stroke, myocardial infarction, other arterial thromboembolism, and all-cause mortality by 30 days following discharge from the hospital.

Biobanking of samples for future biomarker and mechanistic studies will be available for centers able to participate and collect samples from eligible participants. Samples will be collected at the time of enrollment and after the completion of 30 days of therapy

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥ 18 years

  * PCR-positive COVID-19 infection
  * Hospitalized for two or more days

Exclusion Criteria:

* Pre-existing indication for anticoagulation (e.g., pulmonary embolism or deep vein thrombosis; atrial fibrillation; mechanical cardiac valve)
* Contraindication to antithrombotic therapy (e.g., known bleeding within the last 30 days requiring emergency room presentation or hospitalization; major surgery within 14 days; ischemic stroke, intracranial bleed or neurosurgery within 3 months.
* Platelet count < 50,000/mcL
* Hemoglobin <8 gm/dL
* Renal insufficiency (eGFR < 30 mL/min/1.73 m2)
* Pregnancy
* Prison inmate
* Life expectancy less than 90 days
* Unwilling or unable to provide informed consent/unwilling or unable to complete the study protocol
* Dual antiplatelet therapy that cannot be discontinued
* Concomitant need for strong inducers/inhibitors of p-gp or CYP3A4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1291 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-07-24 (Actual); Study Completion 2022-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Wang, MD, Principal Investigator — Duke University
Locations (121):
- United States (121):
  - Valleywise Health Medical Center, Phoenix, Arizona
  - Dignity Health-St Josephs, Phoenix, Arizona
  - Central Arkansas Veterans Health Care System, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Stanford University School of Medicine, Palo Alto, California
  - UCSF at Zuckerberg San Francisco General Hospital, San Francisco, California
  - New Ananda Medical and Urgent Care, Inc., South El Monte, California
  - Mazur and Statner MD PC, Thousand Oaks, California
  - Torrance Medical Center, Torrance, California
  - Centura Health Porter Adventist Hospital, Denver, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - St. Anthony North Health Campus, Westminster, Colorado
  - Baycare Hospital, Clearwater, Florida
  - Florida Heart Center, Ft. Pierce, Florida
  - University of Florida, Gainesville, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Tallahassee Memorial HealthCare, Tallahassee, Florida
  - James A. Haley Veteran's Hospital, Tampa, Florida
  - BayCare Hospital- Winter Haven, Winter Haven, Florida
  - Emory University, Atlanta, Georgia
  - Medical College of Georgia/Augusta University, Augusta, Georgia
  - Savannah Health Services, LLC DBA Memorial Health University Medical Center, Savannah, Georgia
  - Queens Medical Center, Honolulu, Hawaii
  - Hawaii Pacific Health, Honolulu, Hawaii
  - Snake River Research, PLLC, Idaho Falls, Idaho
  - University of Illinois at Chicago, Chicago, Illinois
  - Cook County Health, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - The University of Chicago Medicine, Chicago, Illinois
  - OSF Little Company of Mary, Evergreen Park, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana University Health Bloomington Hospital, Bloomington, Indiana
  - Lutheran Medical Group, Fort Wayne, Indiana
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - Franciscan Health Michigan City, Michigan City, Indiana
  - Reid Physician Associates, Richmond, Indiana
  - Baptist Health Lexington, Lexington, Kentucky
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Clinic Foundation-Baton Rouge, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Willis-Knighton Physician Network/Tri-State Medical Clinic, Shreveport, Louisiana
  - Maine Medical Center/Maine Medical Partners Adult Hospital Medicine, Portland, Maine
  - Pen Bay Medical Center, Rockport, Maine
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Lifebridge (Sinai Hospital of Baltimore), Baltimore, Maryland
  - Adventist HealthCare Shady Grove Medical Center, Rockville, Maryland
  - Boston University, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Baystate Medical center, Springfield, Massachusetts
  - Bay Regional Medical Center d/b/a/ McLaren Bay Region, Bay City, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Western Michigan University, Kalamazoo, Michigan
  - MidMichigan Medical Center, Midland, Michigan
  - McLaren Macomb, Mount Clemens, Michigan
  - Minneapolis VA Health Care System, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Truman Medical Center, Kansas City, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - St Louis University, St Louis, Missouri
  - Mercury Street Medical Group, Butte, Montana
  - CHI St Elizabeth Hospital, Lincoln, Nebraska
  - Renown Health, Reno, Nevada
  - Dartmouth Hichcock Medical Center, Lebanon, New Hampshire
  - AtlantiCare Regional Medical Center, Atlantic City, New Jersey
  - Hope Tower at Jersey Shore University Medical Center, Neptune City, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Capital Health System, Inc., Trenton, New Jersey
  - Christus St. Vincent Regional Medical Center, Santa Fe, New Mexico
  - NYU Langone Hospital-Brooklyn, Brooklyn, New York
  - Coney Island Hospital, Brooklyn, New York
  - Buffalo General Medical Center, Buffalo, New York
  - Mercy Hospital Buffalo, Buffalo, New York
  - Jamaica Hospital Medical Center, Jamaica, New York
  - New York University Langone Health, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - Westchester Medical Center, Valhalla, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke Medical Center, Durham, North Carolina
  - East Carolina University/Vidant Health, Greenville, North Carolina
  - Wake Med Hospital, Raleigh, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Summa Health, Akron, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Ascension St. John Bartlesville, Tulsa, Oklahoma
  - Ascension St. John Tulsa, Tulsa, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - St. Luke's University Health Network, Easton, Pennsylvania
  - Conemaugh Memorial Medical Center, Johnstown, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Tower Health Medical Group, West Reading, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Monument Health Clinical Research, Rapid City, South Dakota
  - Erlanger Health System, Chattanooga, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Christus St. Elizabeth Hospital, Beaumont, Texas
  - Baylor Scott and White Medical Center- College Station, College Station, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Health Harris Methodist, Fort Worth, Texas
  - University of Texas- Houston, LBJ Hospital, Houston, Texas
  - UT Houston MHH-SW, Houston, Texas
  - UTHouston, Houston, Texas
  - Texas Health Frisco, Plano, Texas
  - Baylor Scott and White-Round Rock, Round Rock, Texas
  - Baylor Scott and White-Temple, Temple, Texas
  - The Woodlands Center For Respiratory & Sleep Research, The Woodlands, Texas
  - CHRISTUS Trinity Clinic Pulmonary Medicine, Tyler, Texas
  - The University of Texas Health Science Center at Tyler, Tyler, Texas
  - UT Health East Texas (Tyler), Tyler, Texas
  - UT Rio Grande Valley, Weslaco, Texas
  - MultiCare Institute for Research & Innovation, Puyallup, Washington
  - UW Medicine Valley Medical Center, Renton, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - CAMC Clinical Trials Center, Charleston, West Virginia
  - West Virginia University Hospital, Morgantown, West Virginia
  - Blood Center of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Santos BC, Flumignan RL, Civile VT, Atallah AN, Nakano LC. Prophylactic anticoagulants for non-hospitalised people with COVID-19. Cochrane Database Syst Rev. 2023 Aug 16;8(8):CD015102. doi: 10.1002/14651858.CD015102.pub2. PMID 37591523
- [Derived] Wang TY, Wahed AS, Morris A, Kreuziger LB, Quigley JG, Lamas GA, Weissman AJ, Lopez-Sendon J, Knudson MM, Siegal DM, Kasthuri RS, Alexander AJ, Wahid L, Atassi B, Miller PJ, Lawson JW, Patel B, Krishnan JA, Shapiro NL, Martin DE, Kindzelski AL, Leifer ES, Joo J, Lyu L, Pennella A, Everett BM, Geraci MW, Anstrom KJ, Ortel TL; ACTIV-4C Study Group. Effect of Thromboprophylaxis on Clinical Outcomes After COVID-19 Hospitalization. Ann Intern Med. 2023 Apr;176(4):515-523. doi: 10.7326/M22-3350. Epub 2023 Mar 21. PMID 36940444

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Apixaban
Started | 607 | 610
Completed | 581 | 578
Not Completed | 26 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Apixaban | Total
Number analyzed (Participants) | 607 | 610 | 1217
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54.1 [44 to 64] | 54.1 [44 to 64] | 54.1 [44 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 303 | 311 | 614
  Male | 304 | 299 | 603
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 103 | 100 | 203
  Not Hispanic or Latino | 484 | 487 | 971
  Unknown or Not Reported | 20 | 23 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 363 | 350 | 713
  Asian | 12 | 10 | 22
  Black or African American | 154 | 168 | 322
  American Indian or Alaska Native | 4 | 6 | 10
  Native Hawaiian or other Pacific Islander | 5 | 2 | 7
  Aboriginal or First Nations | 0 | 0 | 0
  Middle Eastern or North African | 0 | 1 | 1
  More than one race | 3 | 5 | 8
  Other Race | 20 | 23 | 43
  Unknown | 46 | 45 | 91
Region of Enrollment [Number; unit: participants]
  United States | 607 | 610 | 1217
Medical history of Deep Vein Thrombosis (DVT) [Count of Participants; unit: Participants] | 7 | 6 | 13
Medical History of Pulmonary Embolism (PE) [Count of Participants; unit: Participants] | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Composite Outcome of Symptomatic Deep Vein Thrombosis, Pulmonary Embolism, Other Venous Thromboembolism, Ischemic Stroke, Myocardial Infarction, Other Arterial Thromboembolism, and All-cause Mortality as Measured by Hospital Records.
Description: Composite endpoint (CE) of venous and arterial thrombotic complications-including new, symptomatic proximal, or distal DVT of the upper or lower extremities, PE, and new thrombosis of other veins (including cerebral sinus and splanchnic veins), ischemic stroke, myocardial infarction, other arterial thromboembolism (e.g., mesenteric or acute limb ischemia), and all-cause mortality by day 30.
Time Frame: 30 days after hospital discharge
Population: intention-to-treat (ITT) population, including all participants randomized
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Apixaban
Number analyzed (Participants) | 607 | 610
percentage of participants | 2.31 [1.27 to 3.84] | 2.13 [1.14 to 3.62]
Statistical Analysis 1: Comparison: Placebo vs Apixaban; Test type: Superiority; Risk Ratio (RR) = 0.92, 95% CI 2-sided [0.44 to 1.95]

2. Secondary Outcome: The Composite Outcome of All-cause Mortality and the EuroQoL Group 5-Dimension (EQ5D) Index Score.
Description: Composite endpoint of mortality and EQ5D index at Day 30. All mortality events will be considered worse than any possible EQ5D response [QOL&M30]. Death was designated as a score of 0. Scores range from 0 (where 0 is the value of a health state equivalent to dead) to 1 (the value of full health), with higher scores indicating higher health utility.
Time Frame: 30 days after hospital discharge
Population: intention-to-treat (ITT) population, including all participants randomized
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | Apixaban
Number analyzed (Participants) | 607 | 610
score on a scale | 0.93 [0.78 to 1.00] | 0.93 [0.75 to 1.00]
Statistical Analysis 1: Comparison: Placebo vs Apixaban; Test type: Superiority; Risk Ratio (RR) = 1.05, 95% CI 2-sided [0.83 to 1.31]

3. Secondary Outcome: The Composite Outcome of All-cause Mortality and the EQ5D Index Score.
Description: Composite endpoint of mortality and EQ5D index at Day 90. All mortality events will be considered worse than any possible EQ5D response. Death was designated as a score of 0. Scores range from 0 (where 0 is the value of a health state equivalent to dead) to 1 (the value of full health), with higher scores indicating higher health utility.
Time Frame: 90 days after hospital discharge
Population: intention-to-treat (ITT) population, including all participants randomized
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | Apixaban
Number analyzed (Participants) | 607 | 610
score on a scale | 0.94 [0.76 to 1.00] | 0.94 [0.74 to 1.00]
Statistical Analysis 1: Comparison: Placebo vs Apixaban; Test type: Superiority; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.78 to 1.24]

4. Secondary Outcome: The Composite Outcome of Symptomatic Deep Vein Thrombosis, Pulmonary Embolism, Other Venous Thromboembolism, Ischemic Stroke, Myocardial Infarction, Other Arterial Thromboembolism, and All-cause Mortality as Measured by Hospital Records.
Time Frame: 45 days after hospital discharge
Population: intention-to-treat (ITT) population, including all participants randomized
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Apixaban
Number analyzed (Participants) | 607 | 610
percentage of participants | 2.80 [1.64 to 4.44] | 2.46 [1.38 to 4.02]
Statistical Analysis 1: Comparison: Placebo vs Apixaban; Test type: Superiority; Risk Ratio (RR) = 0.88, 95% CI 2-sided [0.44 to 1.74]

5. Secondary Outcome: The Composite Outcome of Symptomatic Deep Vein Thrombosis, Pulmonary Embolism, Other Venous Thromboembolism, Ischemic Stroke, Myocardial Infarction, Other Arterial Thromboembolism, and All-cause Mortality as Measured by Hospital Records.
Time Frame: 90 days after hospital discharge
Population: intention-to-treat (ITT) population, including all participants randomized
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Apixaban
Number analyzed (Participants) | 607 | 610
percentage of participants | 2.80 [1.64 to 4.44] | 3.11 [1.89 to 4.82]
Statistical Analysis 1: Comparison: Placebo vs Apixaban; Test type: Superiority; Risk Ratio (RR) = 1.11, 95% CI 2-sided [0.58 to 2.12]

6. Secondary Outcome: New, Symptomatic VTE (Inclusive of DVT, PE, or Other Venous Thrombosis) for up to 30 Days After Randomization as Measured by Hospital Records.
Time Frame: 30 days after randomization (which occurred at time of hospital discharge)
Population: intention-to-treat (ITT) population, including all participants randomized
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Apixaban
Number analyzed (Participants) | 607 | 610
percentage of participants | 0.82 [0.27 to 1.91] | 0.82 [0.27 to 1.90]
Statistical Analysis 1: Comparison: Placebo vs Apixaban; Test type: Superiority; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.29 to 3.42]

7. Secondary Outcome: New, Symptomatic ATE (Inclusive of Ischemic Stroke, MI, or Peripheral Arterial Thromboembolism) for up to 30 Days After Randomization as Measured by Hospital Records.
Time Frame: 30 days after randomization (which occurred at time of hospital discharge)
Population: intention-to-treat (ITT) population, including all participants randomized
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Apixaban
Number analyzed (Participants) | 607 | 610
percentage of participants | 0.49 [0.10 to 1.44] | 0.16 [0.00 to 0.91]
Statistical Analysis 1: Comparison: Placebo vs Apixaban; Test type: Superiority; Risk Ratio (RR) = 0.33, 95% CI 2-sided [0.03 to 3.18]

8. Other Pre Specified Outcome: Percentage of Participants With All-cause Mortality
Time Frame: 30 days following discharge from hospital
Population: intention-to-treat (ITT) population, including all participants randomized
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Apixaban
Number analyzed (Participants) | 607 | 610
percentage of participants | 1.48 [0.68 to 2.80] | 1.31 [0.57 to 2.57]
Statistical Analysis 1: Comparison: Placebo vs Apixaban; Test type: Superiority; Risk Ratio (RR) = 0.88, 95% CI 2-sided [0.34 to 2.28]

9. Other Pre Specified Outcome: The Incidence of All-cause Rehospitalization for up to 90 Days After Randomization
Time Frame: 90 days following discharge from hospital
Reporting Status: Not Posted

10. Other Pre Specified Outcome: The Individual Domains of EQ5D and the EQ5D Visual Analog Scale for 30 and 90 Days After Randomization
Time Frame: 30 and 90 days following discharge from hospital
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to the 90 day visit
Arm/Group | Apixaban | Placebo
All-Cause Mortality (participants affected / at risk) | 12/610 | 9/607
Serious Adverse Events (participants affected / at risk) | 71/610 | 66/607
Other Adverse Events (participants affected / at risk) | 80/610 | 90/607
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apixaban (N=610) | Placebo (N=607)
ACUTE APPENDICITIS (Infections and infestations) | 1 | 0
ACUTE ASTHMA EXACERBATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ACUTE DIFFUSE MYALGIAS (Musculoskeletal and connective tissue disorders) | 1 | 0
ACUTE REJECTION ON TRANSPLANTED KIDNEY (Immune system disorders) | 1 | 0
ALCOHOL DETOXIFICATION (Surgical and medical procedures) | 1 | 0
APPENDICITIS (Infections and infestations) | 0 | 1
ASTHMA EXACERBATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
ATYPICAL CHEST PAIN (General disorders) | 1 | 0
BILATERAL LOWER EXTREMITY CELLULITIS (Infections and infestations) | 0 | 1
BILATERAL PULMONARY EMBOLI (Respiratory, thoracic and mediastinal disorders) | 1 | 1
BRONCHIOLITIS OBLITERANS ORGANIZING PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 | 1
C. DIFFICILE COLITIS (Infections and infestations) | 0 | 2
CARDIAC ARREST (Cardiac disorders) | 1 | 1
CELLULITIS (Infections and infestations) | 0 | 2
CHEST PAIN (General disorders) | 4 | 1
CHRONIC SYSTOLIC HEART FAILURE (Cardiac disorders) | 1 | 0
COMMUNITY ACQUIRED PNEUMONIA (Infections and infestations) | 0 | 1
COMPLEX MIGRAINES (Nervous system disorders) | 0 | 1
COPD EXACERBATION (Respiratory, thoracic and mediastinal disorders) | 2 | 2
COVID-19 PNEUMONIA (Infections and infestations) | 1 | 1
COVID-19 REINFECTION (Infections and infestations) | 0 | 1
CRUSH INJURY (Injury, poisoning and procedural complications) | 1 | 0
CYSTITIS (Infections and infestations) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 | 2
DIABETIC KETO ACIDOSIS (Metabolism and nutrition disorders) | 3 | 1
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
GASTROINTESTINAL BLEED (Gastrointestinal disorders) | 1 | 1
GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 1 | 0
GENERAL WEAKNESS (General disorders) | 2 | 0
GI BLEED (Gastrointestinal disorders) | 1 | 0
HEADACHES (Nervous system disorders) | 1 | 0
HEMATEMESIS (Gastrointestinal disorders) | 1 | 0
HOSPITAL ACQUIRED PNEUMONIA (Infections and infestations) | 1 | 0
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 0 | 1
LEFT LOWER EXTREMITY DVT (Vascular disorders) | 0 | 1
LLE CELLULITIS (Infections and infestations) | 0 | 1
LLE SUPERFICIAL THROMBOSIS (Vascular disorders) | 0 | 1
MITRAL VALVE REGURGITATION (Cardiac disorders) | 0 | 1
NEW ONSET DIABETES (Metabolism and nutrition disorders) | 1 | 0
NON ST SEGMENT ELEVATION MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1
NON-ST ELEVATED MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 | 0
OSTEOMYELITIS (Infections and infestations) | 1 | 0
PANCREATITIS (Gastrointestinal disorders) | 1 | 0
PNEUMONIA (Infections and infestations) | 5 | 5
POST COVID INFLAMMATORY LUNG DISEASE (Infections and infestations) | 1 | 0
POST COVID-19 SYNDROME (Infections and infestations) | 0 | 1
POST-COVID INFLAMMATORY SYNDROME (Infections and infestations) | 1 | 0
POST-SURGICAL INTRA-ABDOMINAL INFECTION (Infections and infestations) | 0 | 1
PULMONARY EMBOLI (Respiratory, thoracic and mediastinal disorders) | 3 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 2
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
SEIZURE (Nervous system disorders) | 0 | 1
SEPTIC SHOCK (Infections and infestations) | 0 | 1
SIALADENITIS (Infections and infestations) | 1 | 0
SIGMOID DIVERTICULITIS (Infections and infestations) | 0 | 1
SMALL BOWEL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1
ST-SEGMENT ELEVATION MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 0
TENSION PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1
TRANSIENT ISCHEMIC ATTACK (Nervous system disorders) | 1 | 0
TRAUMATIC FOLEY INSERTION (Injury, poisoning and procedural complications) | 0 | 1
ULCERATIVE PROCTITIS (Gastrointestinal disorders) | 0 | 1
UNCONTROLLED DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0
WORSENING ABSCESSES (Infections and infestations) | 0 | 1
WORSENING COLLAGENOUS COLITIS (Gastrointestinal disorders) | 1 | 0
WORSENING COVID-19 INFECTION (Infections and infestations) | 0 | 1
WORSENING COVID-19 PNEUMONIA (Infections and infestations) | 10 | 14
WORSENING INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
WORSENING PATHOLOGICAL FRACTURE OF PELVIS (Musculoskeletal and connective tissue disorders) | 1 | 0
WORSENING PNEUMONIA (Infections and infestations) | 4 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apixaban (N=610) | Placebo (N=607)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0
ABNORMAL BLEEDING (Vascular disorders) | 1 | 0
ACUTE BACTERIAL SINUSITIS (Infections and infestations) | 0 | 1
ACUTE PROSTATITIS (Reproductive system and breast disorders) | 0 | 1
ANEMIA (Blood and lymphatic system disorders) | 1 | 0
ANGIONEUROTIC EDEMA (Skin and subcutaneous tissue disorders) | 1 | 0
ANXIETY (Psychiatric disorders) | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
BALANITIS (Reproductive system and breast disorders) | 1 | 0
BILATERAL KNEE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
BILATERAL LEG EDEMA (General disorders) | 0 | 1
BILATERAL LEG PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
BILATERAL LEG SWELLING (General disorders) | 0 | 1
BILATERAL LOWER EXTREMITY PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
BRADYCARDIA (Cardiac disorders) | 0 | 1
BRONCHITIS (Infections and infestations) | 0 | 1
CELLULITIS (Infections and infestations) | 1 | 0
CELLULITIS OF THE RIGHT LOWER EXTREMITY (Infections and infestations) | 1 | 0
CERVICAL RADICULOPATHY (Nervous system disorders) | 0 | 1
CHEST PAIN (General disorders) | 3 | 2
CHEST TIGHTNESS (General disorders) | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 1
COLITIS (Gastrointestinal disorders) | 0 | 1
COMMUNITY ACQUIRED PNEUMONIA (Infections and infestations) | 1 | 0
COMPLEX MIGRAINES (Nervous system disorders) | 0 | 1
COMPLEX REGIONAL PAIN SYNDROME (Nervous system disorders) | 1 | 0
CONCUSSION (Injury, poisoning and procedural complications) | 0 | 1
COPD EXACERBATION (Respiratory, thoracic and mediastinal disorders) | 3 | 0
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 1 | 1
COVID-19 CHRONIC DYSPNEA (Infections and infestations) | 0 | 1
COVID-19 PNEUMONITIS (Infections and infestations) | 1 | 0
DECONDITIONED MUSCLES (Musculoskeletal and connective tissue disorders) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0
DENTAL PAIN (Gastrointestinal disorders) | 0 | 1
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0
DIARRHEA (Gastrointestinal disorders) | 1 | 0
EDEMA (General disorders) | 0 | 1
ELEVATED D-DIMER (Investigations) | 0 | 4
ELEVATED LIVER ENZYMES (Investigations) | 1 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ESOPHAGEAL SPASM (Gastrointestinal disorders) | 0 | 1
FACIAL DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 1
FALL (Injury, poisoning and procedural complications) | 4 | 2
FAULTY OXYGEN EQUIPMENT (Product Issues) | 0 | 1
GASTROESOPHAGEAL REFLUX (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL REFLUX (Gastrointestinal disorders) | 0 | 1
GOUT (Metabolism and nutrition disorders) | 0 | 1
GROUND LEVEL FALL (Injury, poisoning and procedural complications) | 1 | 0
HAIR LOSS (Skin and subcutaneous tissue disorders) | 1 | 0
HEMATOCHEZIA (Gastrointestinal disorders) | 1 | 1
HEMATOMA (Vascular disorders) | 1 | 0
HEMATURIA (Renal and urinary disorders) | 1 | 1
HEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 3
HORSESHOE TEAR OF RETINA WITHOUT DETACHMENT (Eye disorders) | 0 | 1
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPERTENSION (Vascular disorders) | 1 | 0
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
INFLUENZA (Infections and infestations) | 1 | 0
IRRITABLE BOWL SYNDROME (Gastrointestinal disorders) | 0 | 1
LEFT ARM PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
LEFT LOWER EXTREMITY PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
LEFT PLEURITIC CHEST PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1
LEFT SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LOWER EXTREMITY PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
MILD LEFT SYSTOLIC DYSFUNCTION (Cardiac disorders) | 1 | 0
MOTOR VEHICLE ACCIDENT (Injury, poisoning and procedural complications) | 0 | 2
MOTOR VEHICLE VS PEDESTRIAN (Injury, poisoning and procedural complications) | 1 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1
NON-INTRACTABLE HEADACHE (Nervous system disorders) | 0 | 1
NON-OCCLUSIVE THROMBUS (Vascular disorders) | 0 | 1
OTITIS MEDIA (Infections and infestations) | 1 | 0
PALPITATIONS (Cardiac disorders) | 1 | 0
PAROXYSMAL A-FIB (Cardiac disorders) | 0 | 1
PARTIAL MURAL THROMBUS (Vascular disorders) | 1 | 0
PERIVASCULAR DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 2 | 0
PLEURITIC CHEST PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 2
PNEUMONIA (Infections and infestations) | 2 | 0
POST ACUTE COVID-19 SYMPTOMS (Infections and infestations) | 0 | 1
POST ACUTE COVID-19 SYNDROME (Infections and infestations) | 1 | 1
POWER FLOW PORT EVALUATION (Surgical and medical procedures) | 1 | 0
PRURITIC RASH (Skin and subcutaneous tissue disorders) | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 1 | 0
RENAL CALCULI (Renal and urinary disorders) | 0 | 1
RESOLVING COVID-19 PNEUMONIA (Infections and infestations) | 1 | 0
RHEUMATOID ARTHRITIS FLARE UP (Musculoskeletal and connective tissue disorders) | 0 | 1
RIGHT HAND ABSCESS (Infections and infestations) | 0 | 1
RIGHT KNEE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2
RIGHT LEG PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
RIGHT LOWER EXTREMITY PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0
RIGHT RING FINGER LACERATION (Injury, poisoning and procedural complications) | 1 | 0
RIGHT SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
SEIZURE (Nervous system disorders) | 0 | 1
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 1 | 1
SUBSTERNAL CHEST PAIN (General disorders) | 0 | 1
SUPERFICIAL GUN SHOT WOUND (Injury, poisoning and procedural complications) | 0 | 1
SUPERIOR LABRAL TEAR (Injury, poisoning and procedural complications) | 1 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 1
TELOGEN EFFLUVIUM (Skin and subcutaneous tissue disorders) | 1 | 0
TRIQUETRUM FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
TYPE II NSTEMI (Cardiac disorders) | 0 | 1
UNCONTROLLED DIABETES (Metabolism and nutrition disorders) | 1 | 0
UPPER RESPIRATORY INFECTION (Infections and infestations) | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 2
URINARY TRACT INFECTION (Infections and infestations) | 0 | 3
VASOVAGAL SYNCOPE (Nervous system disorders) | 0 | 1
VIRAL SYNDROME (Infections and infestations) | 0 | 1
WEAKNESS (General disorders) | 1 | 0
WORSENING BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
WORSENING CHEST PAIN (General disorders) | 1 | 1
WORSENING CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 0
WORSENING COVID-19 PNEUMONIA (Infections and infestations) | 3 | 5
WORSENING DENTAL PAIN (Gastrointestinal disorders) | 0 | 1
WORSENING DIABETIC FOOT ULCER (Skin and subcutaneous tissue disorders) | 1 | 0
WORSENING HAND TREMOR (Nervous system disorders) | 1 | 0
WORSENING HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
WORSENING INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
WORSENING MOREL LAVALLEE LESION (Musculoskeletal and connective tissue disorders) | 1 | 0
WORSENING NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1
WORSENING PNEUMONIA (Infections and infestations) | 1 | 5
WORSENING VISION LOSS (Eye disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT04650087/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/87/NCT04650087/SAP_001.pdf